CLINICAL TRIAL: NCT00639782
Title: Thromboembolic Related Complications in a Randomized Trial of Previous and Current Generation Mechanical Valve Prostheses
Brief Title: Prospective Randomized On-X Versus SJM Evaluation Trial
Acronym: PROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: On-X Life Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONXSJM1
Record Dates: First submitted 2008-02-16; First posted 2008-03-20 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Heart Valve Disease
Keywords: thromboembolism; mechanical heart valves; randomized
MeSH Terms: conditions — Heart Valve Diseases; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ONX (Active Comparator): On-X heart Valve Replacement
  Interventions: Device: On-X Heart valve replacement
- SJM (Active Comparator): SJM heart valve replacement
  Interventions: Device: SJM Heart valve replacement

INTERVENTIONS:
Device: On-X Heart valve replacement — On-X Heart valve replacement
  Other Names: On-X Prosthetic Heart Valve
  Arms: ONX
Device: SJM Heart valve replacement — SJM Heart valve replacement
  Other Names: St. Jude Medical Prosthetic Heart Valve
  Arms: SJM

SUMMARY:
The study hypothesizes that rate of thromboembolic complications of the On-X prosthesis is reduced as compared to the SJM prosthesis.

DETAILED DESCRIPTION:
The study is a multi-centre, randomized trial that will sequentially enroll up to 500 eligible patients in each group from up to 10 participating study centres internationally to test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient requires an isolated mitral or isolated aortic valve replacement. (Patients undergoing coronary artery bypass and / or concomitant repair of mitral or tricuspid valves are eligible.)
2. The patient is a candidate for receipt of a mechanical heart valve.
3. The patient (or legal guardian) has signed a study-specific informed consent form agreeing to the randomization, data collection and follow-up requirements.
4. The patient can be having a re-operative procedure, so long as the previous prosthetic valve is explanted and the patient does not become a double valve implantation patient.

Exclusion Criteria:

1. The patient is not a candidate to receive a mechanical heart valve.
2. The patient already has a prosthetic valve other than the valve(s) being replaced at this time.
3. The patient requires a tricuspid valve replacement.
4. The patient is enrolled in another investigative study or trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 857 (Actual)
Dates: Start 2003-07; Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Thromboembolisms | 5 years
  Frequency of occurrence for thromboembolic events, either major or reversible, as a function of valve type.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jamieson, MD, Principal Investigator — Vancouver Coastal Health Research Institute
Locations (28):
- United States (7):
  - Southern California Permanente Medical Group, Los Angeles, California
  - Kaiser Foundation Hospital, Honolulu, Hawaii
  - Washington University - St Louis, St Louis, Missouri
  - Christian Hospital Northeast, St Louis, Missouri
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia
- Canada (5):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Heart Institute, Victoria, British Columbia
  - Horizon New Brunswick Heart Centre, Saint John, New Brunswick
  - Jewish General Hospital, Montreal, Quebec
- Germany (4):
  - Universitats-Herzzentrum Bad Krozingen, Freiburg im Breisgau
  - Universitats-Herzzentrum Freiburg - Medical Center, Freiburg im Breisgau
  - Universitats Klinik Jena, Jena
  - Universitat Klinik Tübingen, Tübingen
- India (7):
  - Sri Bachubahi Dayabhai Mehta Mahavir Heart Institute, Surat, Gujarat
  - Shri Jaya Deva Institute of Cardiovascular Sciences, Bangalore, Karnataka
  - Hero Dayanand Medical College and Hospitals, Ludhiana, Punjab
  - Apollo Hospital Chennai, Chennai, Tamil Nadu
  - Frontier Lifeline Hospital, Chennai, Tamil Nadu
  - Apollo Multispecialty Hospitals, Madurai, Tamil Nadu
  - Banaras Hindu University, Varanasi, Uttar Pradesh
- Erasmus Medical Center, Rotterdam, Netherlands
- University of Bergen, Bergen, Norway
- Groote Schuur Hospital, Cape Town, South Africa
- Sahlgrenska University Hospital, Gothenburg, Sweden